CLINICAL TRIAL: NCT06830421
Title: Age-adjusted High-dose Chemotherapy Followed by Autologous Stem Cell Transplantation or Conventional Chemotherapy With R-MP as First-line Treatment in Elderly Primary CNS Lymphoma Patients - a Randomized Phase III Trial
Brief Title: Adjusted High-dose Chemotherapy With Autologous Stem Cell Transplant vs. Conventional Immunochemotherapy in Elderly PCNSL Patients
Acronym: PRIMA-CNS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); University Hospital Tuebingen (Other); Heinrich-Heine University, Duesseldorf (Other); Klinikum Stuttgart (Other); University of Kaiserslautern (Other); University Hospital Munich (Other); University Hospital Regensburg (Other)
Responsible Party: Principal Investigator, Elisabeth Schorb, Principal Investigator, University Hospital Freiburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P003077; 2020-001181-10 (EudraCT Number); DRKS00024085 (Registry Identifier: German Clinical Trials Registry)
Record Dates: First submitted 2023-06-05; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-10

CONDITIONS: Primary Central Nervous System Lymphoma
Keywords: Primary central nervous system lymphoma; HD-chemotherapy followed by autologous stem cell transplantation; Age-adjusted HCT-ASCT; First-line treatment in elderly PCNSL patients; HD-MTX induction

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, open-label, multicenter phase III trial with 2 parallel arms investigating a more intensive, shorter treatment with 2 cycles of MARTA (rituximab, HD-MTX, AraC) followed by HCT with rituximab, busulfan and thiotepa followed by ASCT compared to standard therapy comprising 3 cycles of R-MP followed by procarbazine maintenance for 6 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Active Comparator): Patients will receive 3 cycles (28 days cycle) of R-MP (Rituximab 375 mg/m² i.v. d0,14; MTX 3.5 g/m² i.v. d1,15; Procarbazine 60 mg/m²/d p.o. d2-11) followed by maintenance therapy with Procarbazine 100 mg absolute/d p.o. d1-5 for additional 6 cycles (28 days cycle).
  Interventions: Drug: R-MP and Procarbazine maintenance
- Arm B (Experimental): Patients will receive 2 cycles (21 days cycle) of R-MTX/AraC (Rituximab 375 mg/m² i.v. d0,4; MTX 3.5 g/m² i.v. d1; AraC 2x2 g/m² i.v. d2+d3) followed by consolidating HCT-ASCT with Rituximab 375 mg/m² d-8, Busulfan 3.2 mg/kg/d i.v. d-7 and d-6 and Thiotepa 5 mg/kg/d i.v. d-5 and d-4.
  Interventions: Drug: R-MTX/AraC (MARTA) induction followed by consolidating HCT-ASCT

INTERVENTIONS:
Drug: R-MP and Procarbazine maintenance — Firstline systemic treatment with conventinal immunochemotherapy (3 cycles of Rituximab-MTX-Procarbazine) followed by Procarbazine maintenance
  Arms: Arm A
Drug: R-MTX/AraC (MARTA) induction followed by consolidating HCT-ASCT — Firstline systemic treatment with age-adjusted MTX based induction (2 cycles of Rituximab-Methotrexate-Cytarabin) followed by consolidating aged-adapted high-dose chemotherapy and autologous stem cell transplantation
  Arms: Arm B

SUMMARY:
Most patients being diagnosed with primary diffuse large B-cell lymphoma of the central nervous system (PCNSL) are 60 years or older. Elderly patients with PCNSL have a poor prognosis and there is a great medical need to improve outcome for this vulnerable population. In Germany and many international centres, there are currently two widely used strategies to treat elderly PCNSL patients who are eligible for high-dose methotrexate (HD-MTX) treatment, which have not yet been compared head-to-head. The R-MP regimen has been established by the Cooperative PCNSL Study Group as a "conventional" immunochemotherapy standard treatment for elderly patients with newly diagnosed disease and consists of Rituximab, HD-MTX and Procarbazine followed by maintenance therapy with Procarbazine. In contrast, another recently established protocol also includes HD-MTX-based induction therapy, but followed by consolidating high-dose chemotherapy and autologous stem cell transplantation (HCT-ASCT). This is an overall more intensive, but substantially shorter treatment approach, feasible for elderly patients being considered eligible for a more intensive treatment. The PRIMA-CNS trial aims to compare these two treatment approaches with respect to survival, response rates and toxicity.

DETAILED DESCRIPTION:
Primary diffuse large B-cell lymphoma of the central nervous system (PCNSL) is a rare lymphoma affecting only the central nervous system compartment. PCNSL patients are typically 60 years or older and have poor prognoses. However, there are alternative treatment approaches to consider with the potential to improve medical outcomes for this patient population. The current standard of care in Germany and many international centres for patients 65 and older is treatment with R-MP, comprising rituximab, high-dose methotrexate (HD-MTX) and procarbazine followed by maintenance therapy with procarbazine. An alternative approach comprised of a shorter induction treatment with rituximab, HD-MTX and cytarabine (MARTA) followed by age-adjusted high-dose chemotherapy and autologous stem cell transplantation (HCT-ASCT) was recently shown to be feasible and effective in elderly PCNSL patients considered eligible for high-dose chemotherapy requiring autologous stem cell transplantation. Nevertheless, data evaluating this short duration treatment approach remains scarce, and randomized trials have not yet been published. The objective of the PRIMA-CNS trial is to demonstrate that intensified chemotherapy followed by consolidating HCT-ASCT is superior to conventional chemotherapy with R-MP followed by maintenance with procarbazine in elderly patients with newly diagnosed PCNSL; not only regarding survival and remission after treatment but also regarding standards like quality of life (QOL) and treatment related morbidities. Results of this randomized trial will either change the standard of care to an intense and shorter treatment approach or re-define R-MP as a proven treatment standard. In addition, a geriatric assessement is implemented in this trial with the goal to better define transplant eligibility. If this trial shows the superiority of HCT-ASCT, the investigators will establish an improved treatment standard with increased chances for long-term remission and cure and reduced frequency and length of chemotherapy treatment. Considering the poor prognosis of this patient population, this randomized phase III trial is of great clinical importance to provide patients, the patients' families and care takers with optimal treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Immunocompetent patients with newly-diagnosed primary DLBCL of the central nervous system.
2. Age > 70 years or age 65-70 years if not eligible for more intensive treatment (e.g. OptiMATe trial).
3. Histologically or cytologically assessed diagnosis of B-cell lymphoma by local pathologist.
4. Diagnostic sample obtained by stereotactic or surgical biopsy, cerebrospinal fluid (CSF) cytology examination or vitrectomy.
5. Disease exclusively located in the CNS.
6. At least 1 measurable lesion.
7. Eastern Cooperative Oncology Group (ECOG)-Performance Status (PS) ≤ 2. ECOG PS > 2 accepted if due to PCNSL symptoms.
8. Patients possibly eligible for HCT-ASCT as judged by the treating physician.
9. Written informed consent obtained according to international guidelines and local laws by patient or authorized legal representative in case patient is temporarily legally not competent due to his or her disease.

Additional randomization criteria:

1. Patients eligible for HCT-ASCT defined by the EBL score (at most one of the 3 following conditions may apply: ECOG PS > 1, Barthel Index of activities of daily living (ADL) < 20 and Lachs geriatric screening > 3), improvement of PS after pre-phase treatment or clinical judgement by the treating physician after discussion with the study expert team.
2. No evidence of disease progression after pre-phase treatment.

Exclusion Criteria:

1. Congenital or acquired immunodeficiency including HIV infection and previous organ transplantation.
2. Systemic lymphoma manifestation (outside the CNS).
3. Primary vitreoretinal lymphoma or primary leptomeningeal lymphoma without manifestation in the brain parenchyma or spinal cord.
4. Previous or concurrent malignancies with the exception of surgically cured carcinoma in situ or other kinds of cancer without evidence of disease for at least 5 years.
5. Previous systemic Non-Hodgkin lymphoma at any time.
6. Inadequate renal function (creatinine clearance <60 ml/min).
7. Inadequate bone marrow, cardiac, pulmonary or hepatic function according to investigator´s decision.
8. Active hepatitis B or C disease.
9. Concurrent treatment with other experimental drugs or participation in an interventional clinical trial with administration of study medication within the last thirty days before the start of this study.
10. Third space fluid accumulation >500 ml.
11. Hypersensitivity to study treatment or any component of the formulation.
12. Taking any medications likely to cause interactions with the study medication.
13. Known or persistent abuse of medication, drugs or alcohol.
14. Active COVID-19-infection or non-compliance with the prevailing hygiene measures regarding the COVID-19 pandemic.
15. Patients without legal capacity and who are unable to understand the nature, significance and consequences of the study and without designated legal representative.
16. Previous participation in this trial.
17. Persons who are in a relationship of dependency/employment to the sponsor and/ or investigator.
18. Any familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
19. Fertile patients refusing to use safe contraceptive methods during the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2031-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) between the 2 arms | up to 6 years
  PFS is defined as the time from randomization to disease progression or death of any cause, with censoring at the last date the patient was seen alive and free of disease progression

SECONDARY OUTCOMES:
Overall survival (OS) between the 2 arms | up to 6 years
  OS is defined as time from randomization until death from any cause, with censoring at the last date the patient was seen alive
Event free survival (EFS) between the 2 arms | up to 6 years
  EFS, defined as time from randomization to premature end of treatment (EOT) due to any reason, lymphoma progression or death, whichever occurs first, with censoring at the last date the patient was seen event-free
Remission status after 2 cycles of rituximab-methotrexate-procarbazine (R-MP) (arm A)/2 cycles of R-MTX/cytarabine (AraC) | at RA I: after 8 weeks (Arm A), after 6 weeks (Arm B)
  Remission status after 2 cycles of RMP (arm A) / 2 cycles of R-MTX/AraC will be determined at response assessment (RA) I in both arms and will be divided in complete remission (CR), unconfirmed complete remission (CRu), partial remission (PR), stable disease (SD), progressive disease(PD) according to international PCNSL collaborative group (IPCG) criteria
Remission status after 3 cycles of R-MP (arm A)/consolidating HCT-ASCT (arm B) | at RA II: after 12 weeks
  determined at response assessment (RA) II and will be divided in CR, CRu, PR, SD, PD according to IPCG criteria
Remission status after completion of maintenance treatment (arm A)/6 months follow-up (arm B) | 6 months after RA II
  will be determined 6 months after RA II and will be divided in CR, CRu, PR, SD, PD according to IPCG criteria
Quality of life (EORTC QLQ-C30) | from date of informed consent form (ICF) signature up to 6 years
  EORTC quality of life questionnaire (QLQ)-C30 performed at screening, at RA II /premature EOT and thereafter every 12 months during follow-up
Quality of Life (EORTC-QLQ BN 20) | from date of informed consent form (ICF) signature up to 6 years
  EORTC-QLQ brain neoplasm (BN) 20, performed at screening, at RA II /premature EOT and thereafter every 12 months during follow-up

OTHER OUTCOMES:
Safety: Toxicity | from date of informed consent form (ICF) signature until 30 days after end of treatment
  Incidence of (Serious) adverse events ((S)AE) as assessed by CTCAE v5.0
Safety: Neurotoxicity | from date of informed consent form (ICF) signature up to 6 years
  Results in the following neuropsychological tests: Montreal Cognitive Assessment (MoCA), Trail Making Test A and B, the Rey-Osterrieth-Complex-Figure-Test and a verbal fluency test, performed at screening, RA II / premature EOT and every 12 months during follow-up.
Unplanned hospital admissions | from date of informed consent form (ICF) signature until 30 days after ASCT or 30 days after last administration of investigational medicinal products (IMP)
  Defined as in-patient hospitalization due to SAE from date of informed consent form (ICF) signature until 30 days after ASCT or day 30 after last administration of IMP, whatever occurs first. Each hospitalization will be counted as a single event.
Length of hospital stays | from date of informed consent form (ICF) signature until 30 days after ASCT or day 30 after last administration of IMP
  Measured as number of nights in hospital due to SAE as defined above, i.e. hospital stays from date of ICF signature until 30 days after ASCT or day 30 after last administration of IMP, whatever occurs first.

CONTACTS AND LOCATIONS:
Locations (35):
- Germany (35):
  - University Hospital Freiburg, Department Medicine I, Hematology, oncology and stem cell transplantation, Freiburg im Breisgau, Baden-Wurttemberg
  - Klinikum Stuttgart, Clinic of Hematology, Oncology and Palliative Care, Stuttgart Cancer Center / Tumor Center Eva Mayr-Stihl, Stuttgart, Baden-Wurttemberg
  - University Hospital Aachen, Aachen
  - University Hospital Augsburg, Augsburg
  - Helios Klinikum Berlin-Buch, Berlin
  - University Hospital Berlin, Berlin
  - Evangelisches Klinikum Bethel, Bielefeld
  - Universitätsklinikum Knappschaftskrankenhaus Bochum GmbH, Bochum
  - Städtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Klinikum Bremen-Mitte gGmbH, Bremen
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitätsklinikum Köln, Cologne
  - Carl Gustav Carus Universitätsklinikum Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Essen, Essen
  - Klinikum der Johann-Wolfgang-Goethe-Universität, Frankfurt
  - Universitätsmedizin Göttingen Georg-August-Universität, Göttingen
  - Universitätsklinikum Halle (Saale), Halle
  - Universitätsklinikum des Saarlandes Homburg, Homburg
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - Universitätsklinkum Schleswig-Holstein, Campus Kiel, Kiel
  - Gemeinschaftsklinikum Mittelrhein gGmbH - Koblenz Ev. Stift St. Martin, Koblenz
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Klinikum rechts der Isar TU München, München
  - Universitätsklinikum Münster, Münster
  - Universitätsklinik der Paracelsus Medizinischen Privatuniversität, Nuremberg
  - Pius-Hospital Oldenburg, Oldenburg
  - Klinikum Oldenburg gGmbh, Oldenburg in Holstein
  - Universitätsklinikum Regensburg, Regensburg
  - Universitätsmedizin Rostock, Rostock
  - Universtitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Schwarzwald-Baar-Klinikum Villingen-Schwenningen, Villingen-Schwenningen

IPD SHARING:
Plan to Share IPD: Yes
Publication of study protocol and publication of study results
Supporting Information: Study Protocol
Time Frame: year 2023 and after completion of study
Access Criteria: Isbell LK et al. Age-adjusted high-dose chemotherapy followed by autologous stem cell transplantation or conventional chemotherapy with R-MP as first-line treatment in elderly primary CNS lymphoma patients - the randomized phase III PRIMA-CNS trial. BMC Cancer. 2023 Aug 18;23(1):767.
  doi: 10.1186/s12885-023-11193-7. PMID: 37596517; PMCID: PMC10436648.
URL: https://bmccancer.biomedcentral.com/articles/10.1186/s12885-023-11193-7

REFERENCES:
- [Background] Schorb E, Isbell LK, Kerkhoff A, Mathas S, Braulke F, Egerer G, Roth A, Schliffke S, Borchmann P, Brunnberg U, Kroschinsky F, Mohle R, Rank A, Wellnitz D, Kasenda B, Pospiech L, Wendler J, Scherer F, Deckert M, Henkes E, von Gottberg P, Gmehlin D, Backenstrass M, Jensch A, Burger-Martin E, Grishina O, Fricker H, Malenica N, Orban A, Duyster J, Ihorst G, Finke J, Illerhaus G. High-dose chemotherapy and autologous haematopoietic stem-cell transplantation in older, fit patients with primary diffuse large B-cell CNS lymphoma (MARTA): a single-arm, phase 2 trial. Lancet Haematol. 2024 Mar;11(3):e196-e205. doi: 10.1016/S2352-3026(23)00371-X. Epub 2024 Jan 29. PMID 38301670
- [Background] Mendez JS, Ostrom QT, Gittleman H, Kruchko C, DeAngelis LM, Barnholtz-Sloan JS, Grommes C. The elderly left behind-changes in survival trends of primary central nervous system lymphoma over the past 4 decades. Neuro Oncol. 2018 Apr 9;20(5):687-694. doi: 10.1093/neuonc/nox187. PMID 29036697
- [Background] Houillier C, Soussain C, Ghesquieres H, Soubeyran P, Chinot O, Taillandier L, Lamy T, Choquet S, Ahle G, Damaj G, Agape P, Molucon-Chabrot C, Amiel A, Delwail V, Fabbro M, Jardin F, Chauchet A, Moles-Moreau MP, Morschhauser F, Casasnovas O, Gressin R, Fornecker LM, Abraham J, Marolleau JP, Tempescul A, Campello C, Colin P, Tamburini J, Laribi K, Serrier C, Haioun C, Chebrek S, Schmitt A, Blonski M, Houot R, Boyle E, Bay JO, Oberic L, Tabouret E, Waultier A, Martin-Duverneuil N, Touitou V, Cassoux N, Kas A, Mokhtari K, Charlotte F, Alentorn A, Feuvret L, Le Garff-Tavernier M, Costopoulos M, Mathon B, Peyre M, Delgadillo D, Douzane H, Genet D, Aidaoui B, Hoang-Xuan K, Gyan E. Management and outcome of primary CNS lymphoma in the modern era: An LOC network study. Neurology. 2020 Mar 10;94(10):e1027-e1039. doi: 10.1212/WNL.0000000000008900. Epub 2020 Jan 6. PMID 31907289
- [Background] Schorb E, Fox CP, Kasenda B, Linton K, Martinez-Calle N, Calimeri T, Ninkovic S, Eyre TA, Cummin T, Smith J, Yallop D, De Marco B, Krampera M, Trefz S, Orsucci L, Fabbri A, Illerhaus G, Cwynarski K, Ferreri AJM. Induction therapy with the MATRix regimen in patients with newly diagnosed primary diffuse large B-cell lymphoma of the central nervous system - an international study of feasibility and efficacy in routine clinical practice. Br J Haematol. 2020 Jun;189(5):879-887. doi: 10.1111/bjh.16451. Epub 2020 Jan 29. PMID 31997308
- [Background] Olivier G, Clavert A, Lacotte-Thierry L, Gardembas M, Escoffre-Barbe M, Brion A, Cumin I, Legouffe E, Solal-Celigny P, Chabin M, Ingrand P, Colombat P, Delwail V. A phase 1 dose escalation study of idarubicin combined with methotrexate, vindesine, and prednisolone for untreated elderly patients with primary central nervous system lymphoma. The GOELAMS LCP 99 trial. Am J Hematol. 2014 Nov;89(11):1024-9. doi: 10.1002/ajh.23812. Epub 2014 Aug 27. PMID 25052698
- [Background] Ferreri AJ, Cwynarski K, Pulczynski E, Ponzoni M, Deckert M, Politi LS, Torri V, Fox CP, Rosee PL, Schorb E, Ambrosetti A, Roth A, Hemmaway C, Ferrari A, Linton KM, Ruda R, Binder M, Pukrop T, Balzarotti M, Fabbri A, Johnson P, Gorlov JS, Hess G, Panse J, Pisani F, Tucci A, Stilgenbauer S, Hertenstein B, Keller U, Krause SW, Levis A, Schmoll HJ, Cavalli F, Finke J, Reni M, Zucca E, Illerhaus G; International Extranodal Lymphoma Study Group (IELSG). Chemoimmunotherapy with methotrexate, cytarabine, thiotepa, and rituximab (MATRix regimen) in patients with primary CNS lymphoma: results of the first randomisation of the International Extranodal Lymphoma Study Group-32 (IELSG32) phase 2 trial. Lancet Haematol. 2016 May;3(5):e217-27. doi: 10.1016/S2352-3026(16)00036-3. Epub 2016 Apr 6. PMID 27132696
- [Background] Ferreri AJM, Cwynarski K, Pulczynski E, Fox CP, Schorb E, La Rosee P, Binder M, Fabbri A, Torri V, Minacapelli E, Falautano M, Ilariucci F, Ambrosetti A, Roth A, Hemmaway C, Johnson P, Linton KM, Pukrop T, Sonderskov Gorlov J, Balzarotti M, Hess G, Keller U, Stilgenbauer S, Panse J, Tucci A, Orsucci L, Pisani F, Levis A, Krause SW, Schmoll HJ, Hertenstein B, Rummel M, Smith J, Pfreundschuh M, Cabras G, Angrilli F, Ponzoni M, Deckert M, Politi LS, Finke J, Reni M, Cavalli F, Zucca E, Illerhaus G; International Extranodal Lymphoma Study Group (IELSG). Whole-brain radiotherapy or autologous stem-cell transplantation as consolidation strategies after high-dose methotrexate-based chemoimmunotherapy in patients with primary CNS lymphoma: results of the second randomisation of the International Extranodal Lymphoma Study Group-32 phase 2 trial. Lancet Haematol. 2017 Nov;4(11):e510-e523. doi: 10.1016/S2352-3026(17)30174-6. Epub 2017 Oct 17. PMID 29054815
- [Background] Fritsch K, Kasenda B, Schorb E, Hau P, Bloehdorn J, Mohle R, Low S, Binder M, Atta J, Keller U, Wolf HH, Krause SW, Hess G, Naumann R, Sasse S, Hirt C, Lamprecht M, Martens U, Morgner A, Panse J, Frickhofen N, Roth A, Hader C, Deckert M, Fricker H, Ihorst G, Finke J, Illerhaus G. High-dose methotrexate-based immuno-chemotherapy for elderly primary CNS lymphoma patients (PRIMAIN study). Leukemia. 2017 Apr;31(4):846-852. doi: 10.1038/leu.2016.334. Epub 2016 Nov 15. PMID 27843136
- [Background] Schorb E, Kasenda B, Ihorst G, Scherer F, Wendler J, Isbell L, Fricker H, Finke J, Illerhaus G. High-dose chemotherapy and autologous stem cell transplant in elderly patients with primary CNS lymphoma: a pilot study. Blood Adv. 2020 Jul 28;4(14):3378-3381. doi: 10.1182/bloodadvances.2020002064. PMID 32722778
- [Background] Schorb E, Finke J, Ihorst G, Kasenda B, Fricker H, Illerhaus G. Age-adjusted high-dose chemotherapy and autologous stem cell transplant in elderly and fit primary CNS lymphoma patients. BMC Cancer. 2019 Mar 29;19(1):287. doi: 10.1186/s12885-019-5473-z. PMID 30925912
- [Background] Omuro A, Chinot O, Taillandier L, Ghesquieres H, Soussain C, Delwail V, Lamy T, Gressin R, Choquet S, Soubeyran P, Huchet A, Benouaich-Amiel A, Lebouvier-Sadot S, Gyan E, Touitou V, Barrie M, del Rio MS, Gonzalez-Aguilar A, Houillier C, Delgadillo D, Lacomblez L, Tanguy ML, Hoang-Xuan K. Methotrexate and temozolomide versus methotrexate, procarbazine, vincristine, and cytarabine for primary CNS lymphoma in an elderly population: an intergroup ANOCEF-GOELAMS randomised phase 2 trial. Lancet Haematol. 2015 Jun;2(6):e251-9. doi: 10.1016/S2352-3026(15)00074-5. Epub 2015 Jun 3. PMID 26688235
- [Background] Wendler J, Fox CP, Valk E, Steinheber C, Fricker H, Isbell LK, Neumaier S, Okosun J, Scherer F, Ihorst G, Cwynarski K, Schorb E, Illerhaus G. Optimizing MATRix as remission induction in PCNSL: de-escalated induction treatment in newly diagnosed primary CNS lymphoma. BMC Cancer. 2022 Sep 10;22(1):971. doi: 10.1186/s12885-022-09723-w. PMID 36088292
- [Background] Farhi J, Laribi K, Orvain C, Hamel JF, Mercier M, Sutra Del Galy A, Clavert A, Rousselet MC, Tanguy-Schmidt A, Hunault-Berger M, Moles-Moreau MP. Impact of front line relative dose intensity for methotrexate and comorbidities in immunocompetent elderly patients with primary central nervous system lymphoma. Ann Hematol. 2018 Dec;97(12):2391-2401. doi: 10.1007/s00277-018-3468-5. Epub 2018 Aug 8. PMID 30091022
- [Background] Martinez-Calle N, Isbell LK, Cwynarski K, Schorb E. Advances in treatment of elderly primary central nervous system lymphoma. Br J Haematol. 2022 Feb;196(3):473-487. doi: 10.1111/bjh.17799. Epub 2021 Aug 26. PMID 34448202
- [Background] Schorb E, Isbell LK, Illerhaus G, Ihorst G, Meerpohl JJ, Grummich K, Nagavci B, Schmucker C. Treatment Regimens for Immunocompetent Elderly Patients with Primary Central Nervous System Lymphoma: A Scoping Review. Cancers (Basel). 2021 Aug 24;13(17):4268. doi: 10.3390/cancers13174268. PMID 34503078